CLINICAL TRIAL: NCT06769750
Title: Is the Variability of the Perfusion Index Predictive of Post-spinal Hypotension in Parturients Undergoing Scheduled Cesarean Section
Brief Title: Variability of Perfusion Index to Predict Hypotension
Acronym: IP-HYPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP240165
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Post-spinal Hypotension
Keywords: Spinal anesthesia; Scheduled caesarean section; Parturientes; Post-anaesthetic hypotension; Hypotension prediction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- passive leg-lift (Experimental): A transthoracic cardiac echocardiogram will be performed with measurement of the sub-aortic time-velocity integral, and the same measurement will be performed 1 min after a passive leg-lift to see if this maneuver significantly increases systolic ejection volume. The perfusion index (PI) value and arterial pressure will be measured at each of these manoeuvres. The same data will be collected one minute after return to the initial position. Thereafter, PI and arterial pressure will be recorded every two minutes until the newborn is delivered.
  Interventions: Other: leg-lift maneuver

INTERVENTIONS:
Other: leg-lift maneuver — Patients will be monitored as usual using an SpO2 sensor placed on the index finger of the limb contralateral to the pressure cuff, giving the PI value, a tensiometer taking blood pressure (systolic, diastolic and mean) every 2 minutes, and an ECG.
  A transthoracic cardiac echocardiogram will be performed with measurement of the sub-aortic time-velocity integral, and the same measurement will be performed 1 min after a passive leg-lift to see if this maneuver significantly increases systolic ejection volume. The PI value and blood pressure will be measured at each of these maneuvers.
Other: leg-lift maneuver — The perfusion index (PI) value and arterial pressure will be measured at each of manoeuvre

SUMMARY:
About one-third of deliveries are performed by cesarean section, and this rate is increasing. The standard anesthetic technique for this procedure is spinal anesthesia (SA), which is associated with hypotension in nearly 70% of cases . The mechanism is a sympatholysis leading to a drop in systemic vascular resistance and cardiac output, which can be aggravated by relative hypovolemia. This hypotension is responsible for maternal dizziness, nausea, and vomiting, as well as fetal acidosis, and in extreme cases, fetal circulatory insufficiency.

Currently, it is recommended to prevent post-spinal hypotension through a strategy combining co-loading with fluids and the administration of vasopressors in all patients. However, this non-individualized strategy is not always effective in preventing hypotension and may even be harmful to the mother in cases of excessive fluid administration.

Current guidelines for perioperative fluid management in elective surgery advocate for an individualized approach based on preoperative assessment of preload dependence through cardiac output monitoring. Correcting this relative hypovolemia helps maintain an appropriate blood pressure for the patient's needs.

In parturients, we have shown that evaluating preload dependence by measuring the variation in the time-velocity integral under the aorta (ΔTVI) using cardiac ultrasound before and after a passive leg raising test (PLR) can predict post-spinal hypotension with good sensitivity and specificity. We obtained comparable results using monitoring of the variation in stroke volume by the Clearsight™ system (Edwards Lifesciences, Irvine, California, US), before and after PLR .

However, these technologies have limitations: availability of equipment, cost, operator expertise, and patient echogenicity in the case of ultrasound. Using a non-invasive, simple, and accessible method for monitoring preload dependence that can be used by an untrained operator would help easily identify patients at higher risk for post-spinal hypotension, enabling individualized management.

The main objective of our study is to evaluate the ability of ΔIPELJP to predict post-rachianesthesia hypotension in parturients scheduled for a cesarean section.

DETAILED DESCRIPTION:
This is a prospective, monocentric study carried out at the level 3 maternity unit of Marseille's Hôpital Nord Patients will be monitored as usual using an SpO2 sensor placed on the index finger of the limb contralateral to the blood pressure cuff, giving the PI value, a blood pressure monitor taking blood pressure (systolic, diastolic and mean) every 2 minutes, and an ECG.

A transthoracic cardiac echocardiogram will be performed with measurement of the sub-aortic time-velocity integral, and the same measurement will be taken 1 min after a passive leg-lift to see whether this maneuver significantly increases systolic ejection volume. The PI value and arterial pressure will be measured at each of these manoeuvres. The same data will be collected one minute after return to the initial position. Thereafter, PI and arterial pressure will be recorded every two minutes until the newborn is delivered.

The pH of the newborn's cord blood is systematically recorded.

ELIGIBILITY:
Inclusion Criteria:

* Parturient women
* With a term of more than 34 weeks' amenorrhea (SA)
* Requiring a scheduled caesarean section under spinal anaesthesia at the maternity ward of the Hôpital Nord de Marseille (AP-HM).
* Patients affiliated to a Social Security System

Exclusion Criteria:

* Urgent caesarean section
* Contraindication to perimedullary anesthesia
* Clinical features likely to distort the plethysmographic signal: scleroderma, Raynaud's syndrome, nail pathology, etc.
* Presence of anti-hypertensive treatment
* Cardiac arrhythmia
* Anesthetist not trained in transthoracic cardiac echography
* Refusal to participate in the study
* Guardianship or curatorship, safeguard of justice
* Instable Perfusion Index Signal

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
ΔIPELJP | at the time of cesarean section
  This value will be calculated by subtracting the PI one minute after the passive leg lift from the resting value measured one minute before he passive leg lift was performed.

SECONDARY OUTCOMES:
Incidence of hypotension after rachianesthesia | At the time of cesarean delivery
  Defined as a fall in systolic blood pressure of more than 20% between the resting value before lifting the passive leg and the performance of rachi anesthesia, until delivery of the newborn.
- The delta of PI between PI before spinal anaesthesia and minimum and maximum PI values after spinal anaesthesia and until delivery of the newborn, | At the time of cesarean delivery
  PI will be recorded every minute.
The correlation between ΔIPELJP and ΔITVELJP | Before spinal anaesthesia
Relationship between basal PI and ΔIPELJP to individualize groups at risk of developing hypotension | At the time of cesarean delivery
Correlation between fetal pH value at cord and relationship with initial PI value, PI variation and ΔITVELJP | At delivery
Maximum doses of norepinephrine in mg/h from the time of rachi anesthesia to delivery of the neonate | At delivery
-Cumulative doses of noradrenaline in mg from rachi anesthesia to neonatal delivery | At delivery

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Department of Anesthesia and Intensive Care, Perioperative Medicine, Hôpital Nord,, Marseille, Marseilles
  - Hôpital Nord, Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruscagnin C, Shi R, Rosalba D, Fouque G, Hagry J, Lai C, Donadello K, Pham T, Teboul JL, Monnet X. Testing preload responsiveness by the tidal volume challenge assessed by the photoplethysmographic perfusion index. Crit Care. 2024 Sep 16;28(1):305. doi: 10.1186/s13054-024-05085-w. PMID 39285430
- [Background] Duclos G, Granier S, Hili A, Blanc J, Einav S, Leone M, Zieleskiewicz L. Performance of non-invasive stroke volume variation during passive leg raising as a predictor of hypotension following induction of spinal anesthesia for elective cesarean delivery: a single cohort study. Int J Obstet Anesth. 2022 May;50:103251. doi: 10.1016/j.ijoa.2021.103251. Epub 2021 Dec 30. PMID 35074676
- [Background] Duggappa DR, Lokesh M, Dixit A, Paul R, Raghavendra Rao RS, Prabha P. Perfusion index as a predictor of hypotension following spinal anaesthesia in lower segment caesarean section. Indian J Anaesth. 2017 Aug;61(8):649-654. doi: 10.4103/ija.IJA_429_16. PMID 28890560
- [Background] Beurton A, Gavelli F, Teboul JL, De Vita N, Monnet X. Changes in the Plethysmographic Perfusion Index During an End-Expiratory Occlusion Detect a Positive Passive Leg Raising Test. Crit Care Med. 2021 Feb 1;49(2):e151-e160. doi: 10.1097/CCM.0000000000004768. PMID 33332814
- [Background] Toyama S, Kakumoto M, Morioka M, Matsuoka K, Omatsu H, Tagaito Y, Numai T, Shimoyama M. Perfusion index derived from a pulse oximeter can predict the incidence of hypotension during spinal anaesthesia for Caesarean delivery. Br J Anaesth. 2013 Aug;111(2):235-41. doi: 10.1093/bja/aet058. Epub 2013 Mar 21. PMID 23518802